CLINICAL TRIAL: NCT05076149
Title: A Phase 3, Randomized, Double-blind, Controlled Study Evaluating the Efficacy and Safety of VX-121 Combination Therapy in Subjects With Cystic Fibrosis Who Are Homozygous for F508del, Heterozygous for F508del and a Gating (F/G) or Residual Function (F/RF) Mutation, or Have At Least 1 Other Triple Combination Responsive CFTR Mutation and No F508del Mutation
Brief Title: A Study of VX-121 Combination Therapy in Participants With Cystic Fibrosis (CF) Who Are Homozygous for F508del, Heterozygous for F508del and a Gating (F/G) or Residual Function (F/RF) Mutation, or Have At Least 1 Other Triple Combination Responsive (TCR) CFTR Mutation and No F508del Mutation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX20-121-103; 2021-000694-85 (EudraCT Number)
Record Dates: First submitted 2021-09-29; First posted 2021-10-13 (Actual); Results first posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-05

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — elexacaftor, ivacaftor, tezacaftor drug combination; ivacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ELX/TEZ/IVA (Active Comparator): Following elexacftor/tezacaftor/ivacaftor (ELX/TEZ/IVA) run-in period of 4 weeks, participants received ELX 200 milligram (mg) once daily (qd) /TEZ 100 mg qd/IVA 150 mg every 12 hours (q12h) in the treatment period for 52 weeks.
  Interventions: Drug: ELX/TEZ/IVA; Drug: IVA; Drug: Placebo (matched to VX-121/TEZ/D-IVA)
- VX-121/TEZ/D-IVA (Experimental): Following ELX/TEZ/IVA run-in period of 4 weeks, participants received VX-121 20 mg qd/TEZ 100 mg qd/D-IVA 250 mg qd in the treatment period for 52 weeks.
  Interventions: Drug: VX-121/TEZ/D-IVA; Drug: Placebo (matched to ELX/TEZ/IVA); Drug: Placebo (matched to IVA)

INTERVENTIONS:
Drug: VX-121/TEZ/D-IVA — Fixed-dose combination tablets for oral administration.
  Other Names: VX-121/VX-661/CTP-656; VX-121/VX-661/VX-561; VX-121/tezacaftor/deutivacaftor
  Arms: VX-121/TEZ/D-IVA
Drug: ELX/TEZ/IVA — Fixed-dose combination tablets for oral administration.
  Other Names: VX-445/VX-661/VX-770; elexacaftor/tezacaftor/ivacaftor
  Arms: ELX/TEZ/IVA
Drug: IVA — Tablet for oral administration.
  Other Names: VX-770; ivacaftor
  Arms: ELX/TEZ/IVA
Drug: Placebo (matched to VX-121/TEZ/D-IVA) — Placebo matched to VX-121/TEZ/D-IVA for oral administration.
  Arms: ELX/TEZ/IVA
Drug: Placebo (matched to ELX/TEZ/IVA) — Placebo matched to ELX/TEZ/IVA for oral administration.
  Arms: VX-121/TEZ/D-IVA
Drug: Placebo (matched to IVA) — Placebo matched to IVA for oral administration.
  Arms: VX-121/TEZ/D-IVA

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of VX-121/tezacaftor/deutivacaftor (VX-121/TEZ/D-IVA) in CF participants who are homozygous for F508del, heterozygous for F508del and a gating (F/G) or residual function (F/RF) mutation, or have at least 1 other TCR CF transmembrane conductance regulator (CFTR) gene mutation and no F508del mutation.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant has one of the following genotypes:

  * Homozygous for F508del;
  * Heterozygous for F508del and a gating (F/G) mutation;
  * Heterozygous for F508del and a residual function (F/RF) mutation;
  * At least 1 other TCR CFTR gene mutation identified as responsive to ELX/TEZ/IVA and no F508del mutation
* Forced expiratory volume in 1 second (FEV1) value >=40% and <=90% of predicted mean for age, sex, and height for participants currently receiving CFTR protein modulator therapy; FEV1 >=40% and <=80% for participants not currently receiving CFTR protein modulator therapy

Key Exclusion Criteria:

* History of solid organ or hematological transplantation
* Hepatic cirrhosis with portal hypertension, moderate hepatic impairment (Child Pugh Score 7 to 9), or severe hepatic impairment (Child Pugh Score 10 to 15)
* Lung infection with organisms associated with a more rapid decline in pulmonary status
* Pregnant or breast-feeding females

Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 597 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-11-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (170):
- United States (62):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner University of Arizona Medical Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - University of California Davis Medical Center, Sacramento, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - National Jewish Health, Denver, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - Nemours Children's Specialty Care, Jacksonville, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Central Florida Pulmonary Group, PA, Orlando, Florida
  - Nemours Children's Specialty Care, Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital Outpatient Care Center, St. Petersburg, Florida
  - The Emory Clinic at Chantilly, Atlanta, Georgia
  - St. Luke's Cystic Fibrosis Center of Idaho, Boise, Idaho
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana
  - University of Kentucky, Lexington, Kentucky
  - Tulane Medical Center, New Orleans, Louisiana
  - Maine Medical Partners, Portland, Maine
  - Massachusetts General Hospital Cystic Fibrosis Center Clinical Rsearch Center, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Michigan Medicine, Ann Arbor, Michigan
  - Harper University Hospital, Detroit, Michigan
  - Spectrum Health Medical Group Adult Cystic Fibrosis Care Center, Grand Rapids, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - The Children's Mercy Hospital, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Billings Clinic, Billings, Montana
  - Morristown Medical Center, Morristown, New Jersey
  - CF Therapeutics Development Center of Western New York, Buffalo, New York
  - Northwell Health- Long Island Jewish Medical Center, New Hyde Park, New York
  - Columbia University Medical Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Toledo Children's Hospital/Pediatric Pulmonary & Cystic Fibrosis Center, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Santiago Reyes, M.D., Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Prisma Health Richland Campus, Columbia, South Carolina
  - Sanford Children's Speciality Clinic, Sioux Falls, South Dakota
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - Cook Children's Health Care System, Fort Worth, Texas
  - University of Utah - Primary Children's Medical Center, Salt Lake City, Utah
  - Vermont Lung Center, Colchester, Vermont
  - University of Virginia Health System, Charlottesville, Virginia
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Providence Pediatric Pulmonary & Cystic Fibrosis Clinic, Spokane, Washington
  - West Virginia University, Morgantown, West Virginia
  - University Hospital and UW Health Clinics, Madison, Wisconsin
- Australia (10):
  - Royal Prince Alfred Hospital, Camperdown
  - The Prince Charles Hospital, Chermside
  - Alfred Hospital, Melbourne, VIC
  - Institute for Respiratory Health, Nedlands
  - Telethon Kids Institute, Nedlands
  - The Royal Children's Hospital, Parkville, VIC
  - Sydney Children's Hospital, Randwick
  - Mater Adult Hospital, South Brisbane
  - Queensland Children's Hospital, South Brisbane
  - Westmead Hospital, Westmead
- Austria (5):
  - University of Graz, Graz
  - Medizinische Universität Innsbruck, Innsbruck
  - Uniklinikum Salzburg - Universitätsklinik für Pneumologie/Lungenheilkunde, Salzburg
  - Medizinische Universität Wien, Vienna
  - Abteilung fuer Pulmologie Klinikum Wels-Grieskirchen, Wels
- Belgium (5):
  - Cliniques Universitaires de Bruxelles Hopital Erasme, Brussels
  - Universitair Ziekenhuis Brussel - Campus Jette, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven
  - Cliniques Universitaires Saint-Luc, Woluwe-Saint-Lambert
- Canada (9):
  - University of Calgary Medical Clinic of the Foothills Medical Centre, Calgary
  - Stollery Children's Hospital, Edmonton
  - St. Joseph's Health Care London, London
  - Centre Hospitalier de l'Universite de Montreal (CHUM) Hotel-Dieu, Montreal
  - McGill University Health Centre, Glen Site, Montreal Children's Hospital, Montreal
  - Institut Universitaire de Cardiologie et Pneumologie de Quebec - Universite Laval, Québec
  - St. Michael's Hospital, Toronto
  - British Columbia Children's Hospital, Vancouver
  - St. Paul's Hospital, Vancouver
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Juliane Marie Center, Rigshospitalet, Copenhagen
- France (17):
  - Groupe Hospitaler Pellegrin, CHU De Bordeaux, Bordeaux
  - CHU Lyon - Hopital Femme Mere-Enfant, Bron
  - Centre Hospitalier Intercommunal Creteil, Créteil
  - Institut Cœur Poumon, CHU de Lille, Lille
  - Hopital Arnaud de Villeneuve, Montpellier
  - Centre Hospitalier Universitaire De Nantes - G. R. Laennec, Nantes
  - Centre Hospitalier Universitaire (CHU) de Nice - Hopital Pasteur, Nice
  - Hopital Cochin, Paris
  - Hopital Necker, Enfants Malades, Paris
  - Hopital Robert Debre, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre de Perharidy, Roscoff
  - CHU de Rouen - Hopital Charles Nicolle, Rouen Cedex, Seine Maritime
  - Hôpital de Hautepierre, AX5, Strasbourg
  - Hopital Foch (Suresnes), Hopital Foch, Adultes, Suresnes
  - Hopital Bretonneau, Tours
  - Centre hospitalier universitaire de Nancy, Hôpital de Braboi, Vandœuvre-lès-Nancy
- Germany (6):
  - Charite Paediatric Pulmonology Department, Berlin
  - Friedrich-Alexander University of Erlangen-Nuremberg, University Children's Hospital, Erlangen
  - Ruhrlandklinik Westdeutsches Lungenzentrum am Klinikum Essen, Essen
  - Universitatsklinikum Essen (AoR), Kinderklinik III, Abt. fur Pneumologie, Essen
  - Justus-Liebig-Universität Gießen Zentrum für Kinderheilkunde und Jugendmedizin, Giessen
  - Pneumologisches Studienzentrum Muenchen-West, München
- Greece (2):
  - General Hospital of Thessaloniki "Papanikolaou", Pilea Chortiatis
  - General Hospital of Thessaloniki 'Hippokratio', 3rd Pediatrics Department of Aristotle University of Thessaloniki, Thessaloniki
- Hungary (2):
  - National Koranyi Institute for TBC and Pulmonology, Budapest
  - Pulmonology Institute Torokbalint, Törökbálint
- Ireland (7):
  - Cork University Hospital, Cork
  - Children's Health Ireland at Crumlin, Dublin
  - Children's Health Ireland at Tallaght, Dublin
  - Children's University Hospital, Dublin, Dublin
  - St. Vincent's University Hospital, Dublin
  - University Hospital Limerick (Adults), Limerick
  - University Hospital Limerick (Pediatrics), Limerick
- Israel (3):
  - Hadassah Medical Organization, Jerusalem
  - Schneider Children's Medical Center of Israel, Petach Tikvah
  - Sheba Medical Center - The Edmond and Lili Safra Children's Hospital, Tel Litwinsky
- Italy (8):
  - Azienda Ospedaliero Universitaria Ospedale Riuniti, Ancona
  - Azienda Ospedaliero Universitaria Ospedale Pediatrico Meyer, Florence
  - IRCCS Istituto Giannina Gaslini-Ospedale Pediatrico, Genova
  - Fondazione IRCCS Ospedale Maggiore Policlinico, Mangiagalli e Regina Elena, Milan
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Malattie Apparato Respiratorio 2 - Centro Fibrosi Cistica, Orbassano
  - Centro Regionale Fibrosi Cistica, A.O. Ospedale San Carlo, Potenza
  - Azienda Ospedaliera di Verona - Ospedale Civile Maggiore, Verona
- Netherlands (5):
  - Academisch Medisch Centrum (Academic Medical Centre), Amsterdam
  - UMC St. Radboud, Nijmegen
  - Erasmus Medical Center, Rotterdam
  - HagaZiekenhuis van den Haag, The Hague
  - University Medical Center, Utrecht, Department of Pulmonology and Tuberculosis, Utrecht
- New Zealand (4):
  - Greenlane Clinical Centre, Auckland
  - Starship Children's Hospital, Auckland
  - Canterbury Respiratory Research Group, Christchurch Hospital
  - Waikato Hospital, Hamilton
- Norway (2):
  - Haukeland Universitetssjukehus (CF), Bergen
  - Oslo University Hospital, Department of Paediatric Medicine, Oslo
- Poland (3):
  - Pediatric Hospital Polanki named of Maciej Płażyński, Gdansk
  - Institute of Tuberculosis and Lung Diseases, Rabka-Zdrój
  - Klinika Mukowiscydozy IMD Oddozial Chorob Pluc Szpzoz IM. Dzieci WarszaWY, Łomianki
- Sweden (3):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Lund University Skanes Universitetssjukhus, Malmo
  - Karolinska Universitetssjukhuset, Huddinge, Stockholm
- Switzerland (3):
  - Lindenhofspital - Quartier Bleu, Bern
  - Réseau Hospitalier Neuchâtelois, Neuchâtel
  - Kinderspital Zuerich, Zurich
- United Kingdom (12):
  - Birmingham Children's Hospital, Birmingham
  - Royal Papworth Hospital NHS Foundation Trust, Cambridge
  - Clinical Research Facility, Queen Elizabeth University Hospital, Glasgow
  - Leeds General Infirmary, Leeds
  - St. James University Hospital, Leeds
  - King's College Hospital, London
  - Royal Brompton Hospital, London
  - St. Bartholomew's Hospital, London
  - Royal Manchester Children's Hospital, Manchester
  - Wythenshawe Hospital, Manchester
  - All Wales Adult Cystic Fibrosis Centre, University Hospital Llandough, Penarth
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing

REFERENCES:
- [Derived] Keating C, Yonker LM, Vermeulen F, Prais D, Linnemann RW, Trimble A, Kotsimbos T, Mermis J, Braun AT, O'Carroll M, Sutharsan S, Ramsey B, Mall MA, Taylor-Cousar JL, McKone EF, Tullis E, Floreth T, Michelson P, Sosnay PR, Nair N, Zahigian R, Martin H, Ahluwalia N, Lam A, Horsley A; VX20-121-102 Study Group; VX20-121-103 Study Group. Vanzacaftor-tezacaftor-deutivacaftor versus elexacaftor-tezacaftor-ivacaftor in individuals with cystic fibrosis aged 12 years and older (SKYLINE Trials VX20-121-102 and VX20-121-103): results from two randomised, active-controlled, phase 3 trials. Lancet Respir Med. 2025 Mar;13(3):256-271. doi: 10.1016/S2213-2600(24)00411-9. Epub 2025 Jan 2. PMID 39756424
- [Derived] Heneghan M, Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2023 Nov 20;11(11):CD010966. doi: 10.1002/14651858.CD010966.pub4. PMID 37983082

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in cystic fibrosis (CF) participants aged 12 years or older. It was pre-specified in the protocol to combine the data from this study with study VX20-121-102 (NCT05033080) for selected outcome measures.
Pre-assignment Details: A total of 597 participants were enrolled in this study, of which 24 were included in the run-in period but were not dosed in treatment period. Therefore, results are presented for only 573 participants dosed in the treatment period.
Groups:
- ELX/TEZ/IVA: Following elexacaftor/tezacaftor/ivacaftor (ELX/TEZ/IVA) run-in period of 4 weeks, participants received ELX 200 milligram (mg) once daily (qd)/TEZ 100 mg qd/IVA 150 mg every 12 hours (q12h) in the treatment period for 52 weeks.
Period: Overall Study
Arm/Group | ELX/TEZ/IVA | VX-121/TEZ/D-IVA
Started | 289 | 284
Pooled Analysis Set (The Pooled Full Analysis Set (PFAS) included all randomized participants from this study (VX20-121-103) and from Study VX20-121-102 who carry the intended CFTR genotype and received at least 1dose of study drug during the Treatment Period.) | 491 (Out of 491 participants, 289 participants were enrolled from this study and 202 participants were enrolled from VX20-121-102 study.) | 480 (Out of 480 participants, 284 participants were enrolled from this study and 196 participants were enrolled from VX20-121-102 study.)
Completed | 279 | 264
Not Completed | 10 | 20
Not completed — Adverse Event | 3 | 9
Not completed — Withdrawal of consent (not due to AE) | 1 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Commercial drug is available for participant | 0 | 1
Not completed — Other non compliance | 1 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Other | 5 | 4

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug during the treatment Period.
Groups:
- ELX/TEZ/IVA: Following ELX/TEZ/IVA run-in period of 4 weeks, participants received ELX 200 mg qd/TEZ 100 mg qd/IVA 150 mg q12h in the treatment period for 52 weeks.
- Total: Total of all reporting groups
Arm/Group | ELX/TEZ/IVA | VX-121/TEZ/D-IVA | Total
Number analyzed (Participants) | 289 | 284 | 573
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.0 (12.4) | 33.3 (12.6) | 33.7 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 135 | 280
  Male | 144 | 149 | 293
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 261 | 265 | 526
  Not Collected per Local Regulations | 23 | 15 | 38
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 262 | 270 | 532
  Asian | 1 | 1 | 2
  American Indian or Alaska Native | 1 | 0 | 1
  Other | 1 | 1 | 2
  Not Collected per Local Regulations | 23 | 10 | 33
  More than one race | 1 | 2 | 3
Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) [Mean (Standard Deviation); unit: Percentage points] — FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. Population: Here, "Number Analyzed" signifies participants who were evaluable for this study specific baseline measure. This analysis set (N=565) included participants who received the dose and who had a data for this efficacy analysis.
  Percentage points
    number analyzed (Participants) | 286 | 279 | 565
    (all) | 66.4 (14.9) | 67.2 (14.6) | 66.8 (14.7)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Percent Predicted Forced Expiratory Volume in 1second (ppFEV1)
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: From Baseline Through Week 24
Population: The Full Analysis Set (FAS) included all randomized participants who carried the intended CFTR mutation(s) and received at least 1 dose of study drug during the Treatment Period. Here "Overall Number of participants Analyzed" signifies those participants who were evaluated for this specific outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage points
Arm/Group | ELX/TEZ/IVA | VX-121/TEZ/D-IVA
Number analyzed (Participants) | 276 | 268
percentage points | 0.0 [-0.5 to 0.5] | 0.2 [-0.3 to 0.7]
Statistical Analysis 1: Comparison: ELX/TEZ/IVA vs VX-121/TEZ/D-IVA; Test type: Non-Inferiority — The non-inferiority margin represents a clinically acceptable loss of effectiveness that margin preserve at least 50% of the treatment effect of the active control (ELX/TEZ/IVA) compared to placebo, where the treatment effect is estimated by the lower bound of the 95% confidence interval (CI); p < 0.0001, Mixed Models Repeated Measures; LS Mean difference = 0.2, 95% CI 2-sided [-0.5 to 0.9]

2. Secondary Outcome: Absolute Change in Sweat Chloride (SwCl)
Description: Sweat samples were collected using an approved collection device.
Time Frame: From Baseline Through Week 24
Population: FAS. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this specific outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimole per liter (mmol/L)
Arm/Group | ELX/TEZ/IVA | VX-121/TEZ/D-IVA
Number analyzed (Participants) | 276 | 270
millimole per liter (mmol/L) | -2.3 [-3.6 to -0.9] | -5.1 [-6.4 to -3.7]
Statistical Analysis 1: Comparison: ELX/TEZ/IVA vs VX-121/TEZ/D-IVA; Test type: Superiority; p = 0.0034, Mixed Models Repeated Measures; LS Mean difference = -2.8, 95% CI 2-sided [-4.7 to -0.9]

3. Secondary Outcome: Percentage of Participants With SwCl <60 Millimole Per Liter (mmol/L) (Pooled With Data From Study VX20-121-102)
Description: Sweat samples were collected using an approved collection device.
Time Frame: From Baseline Through Week 24
Population: The Pooled Full Analysis Set (PFAS) included all randomized participants from this study (VX20-121-102) and from Study VX20-121-103 who carried the intended CFTR mutation(s) and received at least 1 dose of study drug during the Treatment Period. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this specific outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | ELX/TEZ/IVA | VX-121/TEZ/D-IVA
Number analyzed (Participants) | 479 | 465
percentage of participants | 76.6 | 85.8
Statistical Analysis 1: Comparison: ELX/TEZ/IVA vs VX-121/TEZ/D-IVA; Test type: Other; p < 0.0001, Generalized Estimated Equation Model; Odds Ratio (OR) = 2.21, 95% CI 2-sided [1.55 to 3.16]

4. Secondary Outcome: Percentage of Participants With SwCl <30 mmol/L (Pooled With Data From Study VX20-121-102)
Description: Sweat samples were collected using an approved collection device.
Time Frame: From Baseline Through Week 24
Population: PFAS. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this specific outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | ELX/TEZ/IVA | VX-121/TEZ/D-IVA
Number analyzed (Participants) | 479 | 465
percentage of participants | 22.5 | 30.5
Statistical Analysis 1: Comparison: ELX/TEZ/IVA vs VX-121/TEZ/D-IVA; Test type: Other; p < 0.0001, Generalized Estimated Equation Model; Odds Ratio (OR) = 2.87, 95% CI 2-sided [2.00 to 4.12]

ADVERSE EVENTS:
Time Frame: Day 1 up to Safety follow-up (up to 56 weeks)
Description: Safety set include all participants who received at least 1 dose of study drug during the Treatment Period.
Groups:
- ELX/TEZ/IVA: Following ELX/TEZ/IVA run-in period of 4 weeks, subjects received ELX 200 mg qd /TEZ 100 mg qd/IVA 150 mg q12h in the treatment period for 52 weeks.
Arm/Group | ELX/TEZ/IVA | VX-121/TEZ/D-IVA
All-Cause Mortality (participants affected / at risk) | 0/289 | 0/284
Serious Adverse Events (participants affected / at risk) | 40/289 | 40/284
Other Adverse Events (participants affected / at risk) | 253/289 | 252/284
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ELX/TEZ/IVA (N=289) | VX-121/TEZ/D-IVA (N=284)
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Vision blurred (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 2 | 1
Faecaloma (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
Pancreatic cyst (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 0
Fatty liver alcoholic (Hepatobiliary disorders) | 1 | 0
COVID-19 (Infections and infestations) | 1 | 1
Erysipelas (Infections and infestations) | 0 | 1
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 | 1
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 12 | 18
Influenza (Infections and infestations) | 2 | 4
Lower respiratory tract infection bacterial (Infections and infestations) | 1 | 0
Metapneumovirus pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 6 | 2
Pyelonephritis (Infections and infestations) | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Skull fractured base (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 2
Blood bilirubin increased (Investigations) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 2
Glycosylated haemoglobin increased (Investigations) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Type 3 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Post-traumatic headache (Nervous system disorders) | 0 | 1
Psychomotor hyperactivity (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 1
Device leakage (Product Issues) | 0 | 1
Acute stress disorder (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 2 | 0
Intermenstrual bleeding (Reproductive system and breast disorders) | 1 | 0
Vaginal cyst (Reproductive system and breast disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ELX/TEZ/IVA (N=289) | VX-121/TEZ/D-IVA (N=284)
Abdominal pain (Gastrointestinal disorders) | 23 | 15
Constipation (Gastrointestinal disorders) | 19 | 15
Diarrhoea (Gastrointestinal disorders) | 44 | 37
Nausea (Gastrointestinal disorders) | 13 | 22
Vomiting (Gastrointestinal disorders) | 19 | 12
Fatigue (General disorders) | 30 | 33
Pyrexia (General disorders) | 29 | 28
COVID-19 (Infections and infestations) | 72 | 57
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 85 | 70
Influenza (Infections and infestations) | 14 | 29
Nasopharyngitis (Infections and infestations) | 60 | 57
Sinusitis (Infections and infestations) | 26 | 9
Upper respiratory tract infection (Infections and infestations) | 40 | 55
Viral upper respiratory tract infection (Infections and infestations) | 17 | 20
Alanine aminotransferase increased (Investigations) | 18 | 24
Aspartate aminotransferase increased (Investigations) | 18 | 19
Blood creatine phosphokinase increased (Investigations) | 17 | 24
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 | 14
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 16
Headache (Nervous system disorders) | 41 | 51
Anxiety (Psychiatric disorders) | 6 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 60 | 63
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21 | 11
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 22 | 16
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 23 | 29
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 37 | 45
Productive cough (Respiratory, thoracic and mediastinal disorders) | 19 | 16
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 22 | 16
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 10 | 18
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 29 | 27
Rash (Skin and subcutaneous tissue disorders) | 13 | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-08-19): https://cdn.clinicaltrials.gov/large-docs/49/NCT05076149/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-19): https://cdn.clinicaltrials.gov/large-docs/49/NCT05076149/SAP_001.pdf